CLINICAL TRIAL: NCT00023374
Title: TBTC Study 24: A Non-Comparative Study of the Efficacy of a Largely-Intermittent, Six-Month Tuberculosis Treatment Regimen Among Patients Who Will Not Receive Isoniazid Due to Initial Isoniazid Resistance or Intolerance
Brief Title: TBTC Study 24: Intermittent Treatment of TB With Isoniazid Resistance or Intolerance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Stefan Goldberg, CDC
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDC-NCHSTP-2340; 24
Record Dates: First submitted 2001-09-06; First posted 2001-09-10 (Estimated); Last update posted 2011-08-03 (Estimated); Status verified 2011-06

CONDITIONS: Tuberculosis
Keywords: tuberculosis; TB; isoniazid resistance; isoniazid intolerance; treatment; efficacy; toxicity
MeSH Terms: conditions — Tuberculosis | interventions — Rifampin; Pyrazinamide; Ethambutol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rifampin+PZA+Ethambutol (Experimental): 6 mos of intermittent (2 or 3 times weekly) therapy with REZ
  Interventions: Drug: Rifampin; Drug: Pyrazinamide; Drug: Ethambutol; Drug: REZ

INTERVENTIONS:
Drug: Rifampin — 6mos REZ intermittent
Drug: Pyrazinamide — 6mos REZ intermittent
Drug: Ethambutol — 6mos REZ intermittent
Drug: REZ — Rif+PZA+EMB given 2 or 3 times weekly for 6 months

SUMMARY:
This study is a prospective, open-label, nonrandomized trial using a largely-intermittent, six-month tuberculosis treatment regimen among patients who will not receive isoniazid due to the presence of initial isoniazid resistance or intolerance. Subjects are enrolled after resistance or intolerance to isoniazid has been documented, and are treated for a total of six months (nine months if baseline chest x-ray shows cavitation and 2-month sputum culture is positive) with twice weekly or thrice weekly rifampin, ethambutol, and pyrazinamide.

DETAILED DESCRIPTION:
Primary Objective:

To evaluate the efficacy of a directly-observed, largely-intermittent, six-month regimen of rifampin, pyrazinamide, ethambutol among patients with culture confirmed isoniazid-resistant M. tuberculosis.

Secondary Objectives:

To describe the rate, severity and timing of toxicities and drug intolerances associated with this treatment regimen.

To describe the utility of this regimen among patients who are unable to continue the standard 4-drug regimen due to the development of intolerance to isoniazid

ELIGIBILITY:
Inclusion criteria:

1. Culture-confirmed pulmonary or extrapulmonary tuberculosis due to a strain of M tuberculosis sensitive to rifampin, ethambutol and pyrazinamide based upon specimens (sputum or other pulmonary or extrapulmonary disease site specimens) collected no more than 8 weeks before and no more than 2 weeks after the start of the initial therapy. Susceptibility testing results documenting susceptibility to rifampin and ethambutol must be available at the time of enrollment. Susceptibility results to pyrazinamide may be pending at enrollment as long as pyrazinamide resistance is not known to be present based on prior testing. If pyrazinamide resistance is detected and confirmed (see Study Definitions) the patient will be withdrawn from the study therapy, treatment continued as recommended by the treating physician, and follow-up continued as per the protocol.
2. Decision to discontinue or not use isoniazid for one or both of these following conditions within the first 70 days of therapy:

   * Isoniazid resistant strain (growth in 0.2 mcg/ml or 0.1 mcg/ml of isoniazid on solid or liquid media, respectively)
   * The discontinuation of isoniazid due to intolerance (as judged by the principal investigator - see Study Definitions)
3. For patients enrolled after the start of therapy, documentation of adequate initial regimen as recommended in the CDC/ATS Treatment Guidelines (Appendix 1) is required. There are two means by which this requirement can be met:

   * The standard 4-drug regimen of isoniazid, rifampin, pyrazinamide, and either ethambutol or streptomycin or both.
   * The same regimen with isoniazid excluded for some or all doses in patients with known isoniazid intolerance or tuberculosis due to an isoniazid-resistant strain (i.e., the 3-drug regimen of rifampin, pyrazinamide and either ethambutol or streptomycin or both)
4. A minimum duration of daily treatment as defined by one of two methods:

   * 14 daily doses within 17 days (with at least 10 of the 14 doses directly observed)
   * 14 directly observed doses within 23 days

   Following the minimum daily phase of therapy, adequate pre-enrollment treatment is defined as directly administered therapy given daily, twice weekly, or thrice weekly using CDC/ATS guidelines. Documenting pre-enrollment therapy is accomplished by hospital medical records and/or clinic entries of DOT.
5. Age: 18 years or older
6. Documentation of negative test for human immunodeficiency virus (HIV) infection. Documentation means written copies of HIV laboratory test results. A negative HIV test result within the 6 months prior to enrollment is acceptable.
7. Documentation of study baseline laboratory parameters. Baseline laboratory parameters obtained no more than 2 weeks prior to enrollment and must be within the following limits:

   1. . Amino aspartate transferase (AST) activity less than 3 times upper limit of normal;
   2. . Total bilirubin level less than 2.5 times upper limit of normal;
   3. . Creatinine level less than 2 times upper limit of normal;
   4. . Hemoglobin level of at least 7.0 g/dL;
   5. . Platelet count of at least 50,000 mm3
8. Karnofsky score of at least 60. See Appendix 6 for Karnofsky scoring system.
9. A negative pregnancy test within the past 14 days for women with child-bearing potential, and a willingness to practice an adequate (preferably barrier) method of birth control. In addition, women with child-bearing potential should be offered information concerning sources of contraceptive counseling and services.
10. Informed consent signed by patient and investigator documenting the willingness to use the 3-drug, intermittent regimen is required, in accordance with state law and local IRB requirements. Patients who are unable to provide informed consent due to an inability to comprehend English may be enrolled by providing informed consent by either of two means:

    * the use of a translator to provide a verbal translation of the IRB-approved English version of the consent form; the translator will sign the English form attesting the translation and the patient will sign the IRB-approved translation of the short form
    * the use of a translated consent document, approved by the IRB, that is in the patient's native language.

Exclusion criteria

1. Patients with known treatment-limiting reaction to rifamycins, pyrazinamide, or ethambutol.
2. Diagnosis of silicotuberculosis or tuberculosis of the central nervous system
3. Patients who, during initial therapy with CDC/ATS recommended therapy with isoniazid, rifampin and pyrazinamide plus either ethambutol or streptomycin or both, have received greater than 21 days of treatment with additional drugs with known antituberculosis activity - see Concomitant Medications During Study Phase Therapy.
4. Patients with isoniazid intolerance or isoniazid-resistant tuberculosis who during pre-enrollment therapy have missed a total of two weeks of directly observed therapy doses due to non-compliance.
5. Patients enrolled due to isoniazid intolerance who during pre-enrollment therapy have missed a total of over 4 weeks of directly observed therapy doses for management of drug intolerance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2000-08; Primary Completion 2006-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Combined endpoint of bacteriologic plus clinical failure and relapse within 2 years of completing treatment among patients with isoniazid-resistant tuberculosis and among patients enrolled with intolerance to isoniazid | 30 mos

SECONDARY OUTCOMES:
Occurrence and timing of toxicities and drug intolerances | 6 mos
Time to completion and the frequency of successful completion | 6 mos
Occurrence of acquired resistance | 30 mos
Proportion with documented conversion of 8-week sputum cultures | 8 wks
Bacteriologic failure or relapse in patients with resistance to streptomycin | 30 mos
Bacteriologic failure or relapse among patient with history of prior treatment | 30 mos
Bacteriologic failure or relapse by duration of isoniazid received | 30 mos
Bacteriologic failure or relapse among patients with positive 8-week sputum cultures | 30 mos

CONTACTS AND LOCATIONS:
Overall Officials: Randall Reves, MD, Principal Investigator — Denver Health and Hospitals, Denver CO
Locations (23):
- United States (20):
  - Central Arkansas Veterans Health System, Little Rock, Arkansas
  - LA County/USC Medical Center, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Denver Department of Public Health and Hospitals, Denver, Colorado
  - Washington, D.C. VAMC, Washington D.C., District of Columbia
  - Chicago VA Medical Center (Lakeside), Chicago, Illinois
  - Hines VA Medical Center, Hines, Illinois
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - New Jersey Medical School, Newark, New Jersey
  - New York University School of Medicine, New York, New York
  - Columbia University/Presbyterian Medical Center, New York, New York
  - Harlem Hospital Center, New York, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Nashville VA Medical Center, Nashville, Tennessee
  - University of North Texas Health Science Center, Fort Worth, Texas
  - Thomas Street Clinic, Houston, Texas
  - Audi L. Murphy VA Hospital, San Antonio, Texas
  - Seattle King County Health Department, Seattle, Washington
- Canada (3):
  - University of British Columbia, Vancouver, British Columbia
  - University of Manitoba, Winnipeg, Manitoba
  - Montreal Chest Institute McGill University, Montreal, Quebec

REFERENCES:
- [Derived] Reves R, Heilig CM, Tapy JM, Bozeman L, Kyle RP, Hamilton CD, Bock N, Narita M, Wing D, Hershfield E, Goldberg SV; Tuberculosis Trials Consortium. Intermittent tuberculosis treatment for patients with isoniazid intolerance or drug resistance. Int J Tuberc Lung Dis. 2014 May;18(5):571-80. doi: 10.5588/ijtld.13.0304. PMID 24903795
- [Derived] Funck-Jensen KL, Dalsgaard J, Grove EL, Hvas AM, Kristensen SD. Increased platelet aggregation and turnover in the acute phase of ST-elevation myocardial infarction. Platelets. 2013;24(7):528-37. doi: 10.3109/09537104.2012.738838. Epub 2012 Dec 5. PMID 23216571
- See also: (Click here for more information about the Tuberculosis Trials Consortium(TBTC — http://www.cdc.gov/nchstp/tb/tbtc/